CLINICAL TRIAL: NCT07261501
Title: An Exploratory Research on the Efficacy and Safety of Antibacterial Absorbable Dressing in Chronic Non-healing Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Professor, Head of Wound Healing Center, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Long2025-CW-antibiodegrade
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Wound Heal; Wound Healing Delayed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): On the basis of standard clinical treatment, use of antimicrobial absorbable wound dressing for 3 weeks
  Interventions: Device: antimicrobial absorbable wound dressing
- control group (No Intervention): standard clinical treatment

INTERVENTIONS:
Device: antimicrobial absorbable wound dressing — Perform wound bed preparation per clinical routine protocols . Choose an appropriately sized product based on wound dimensions. Peel open the outer aluminum foil pouch from the hermetically sealed edge; the inner pouch remains sterile and may be placed in a sterile field . If necessary, rinse surgical gloves with powder-free solution before handling the product. The material can be trimmed in either moist or dry conditions. Sterile room-temperature irrigation solution may be used for moistening as needed Place either side of the product against the wound, ensuring complete coverage with slight overhang beyond the wound edge. Re-moisten the product with sterile room-temperature irrigation solution if required . Use an appropriate secondary dressing to maintain adherence and prevent displacement.
  Arms: test group

SUMMARY:
Antimicrobial absorbable wound dressing is a novel polyester-based degradable dressing. Previous preclinical studies have demonstrated promising efficacy, with a 3-week wound area reduction rate of 63.53% in large animal models, outperforming foreign counterparts (49.47%), without significant adverse reactions observed during application. Toxicological risk assessment confirms acceptability, and small animal model studies show no abnormalities in toxicity or sensitization. However, current evidence lacks clinical validation, particularly regarding efficacy and safety in chronic non-healing wounds.

This study integrates modern clinical evaluation methods with chronic wound staging theory to systematically investigate the effectiveness and safety of antimicrobial absorbable wound repair materials in treating chronic non-healing wounds. The research aims to identify optimal indications and provide robust evidence for its clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-80 years
* Wound Type : Chronic non-healing ulcers* with no signs of healing progression for ≥1 week
* Wound Area : 1-35 cm²
* Infection Status : Local infection, contamination, or colonization** as classified by IWII Wound Infection Staging
* Wound Phase : Late necrotic stabilization phase, granulation phase, or epithelial migration phase***
* Consent : Voluntary participation with signed informed consent

Exclusion Criteria:

* Severe Comorbidities : Acute myocardial infarction, heart failure, hepatitis, shock, respiratory failure, or other critical conditions requiring stabilization
* Uncontrolled Diabetes : Fasting blood glucose >15 mmol/L or HbA1c >12%
* Active Wound Hemorrhage : Bleeding precluding standard wound therapy
* Critical Laboratory Values :

Serum albumin <20 g/L Hemoglobin <60 g/L Platelet count <50×10⁹/L

* Systemic Infection : Disseminated/systemic infection requiring antibiotic therapy
* Malignancy : Advanced cancer patients，Current radiotherapy/chemotherapy，Malignant (cancer-related) ulcers
* Untreated Burns : Full-thickness (third-degree) burns without escharotomy
* Active Autoimmune Disease : Flare-up phase of autoimmune disorders
* Pregnancy/Lactation : Pregnant or breastfeeding women
* Allergy : Hypersensitivity to absorbable wound repair materials or polyhexamethylene biguanide hydrochloride
* Non-compliance : Inability to cooperate or psychiatric disorders
* Investigator's Discretion : Any condition deemed to compromise wound healing or study adherence

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Wound Area Reduction Rate at 3 Weeks | Day 21±2
  The 3-week wound area reduction rate (%) is calculated as:
  Reduction Rate (%) = （Baseline Wound Area (D0)-Wound Area Post-Treatment (D21)）/Baseline Wound Area (D0) × 100%

SECONDARY OUTCOMES:
Wound Healing Rate at 3 Weeks | Day 21±2
  The percentage of completely healing wound at 3 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No